CLINICAL TRIAL: NCT00396448
Title: A 2-Year, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study To Evaluate The Long-Term Efficacy And Safety Of CP-945,598 In The Treatment Of Obese Subjects
Brief Title: Effect of 2-year Administration of CP-945,598 on Weight Loss Efficacy and Safety.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5351019
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CP-945,598 Treatment B (Experimental)
  Interventions: Drug: CP-945,598 Treatment B
- CP-945,598 Treatment A (Experimental)
  Interventions: Drug: CP-945,598 Treatment A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-945,598 Treatment B — Subjects receive CP-945,598 plus dietary, physical activity, and behavioral counseling.
  Arms: CP-945,598 Treatment B
Drug: CP-945,598 Treatment A — Subjects receive CP-945,598 plus dietary, physical activity, and behavioral counseling.
  Arms: CP-945,598 Treatment A
Drug: Placebo — Subjects receive placebo plus dietary, physical activity, and behavioral counseling.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the long-term weight loss and safety of CP-945,598 in obese adults

DETAILED DESCRIPTION:
The CP-945,598 program was terminated on November 3, 2008 due to changing regulatory perspectives on the risk/benefit profile of the CB1 class and likely new regulatory requirements for approval. No safety issues were involved in the termination decision.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults with a body mass index > or = 30 kg/m ; > or = 27 kg/m2 for those with obesity-related comorbidities including hypertension and dyslipidemia

Exclusion Criteria:

* Pregnancy
* Diabetes
* Adults with serious or unstable current or past medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1253 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in body weight and proportion of subjects with 5% weight loss | 1 year

SECONDARY OUTCOMES:
Waist circumference, blood lipids and glucose, prevalence of metabolic syndrome, patient reported outcomes, population PK | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (55):
- United States (15):
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Bountiful, Utah
- Argentina (6):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Ramos Mejía, Buenos Aires
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, Villa Carlos Paz, Córdoba Province
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Capital Federal
- Australia (7):
  - Pfizer Investigational Site, Caringbah, New South Wales
  - Pfizer Investigational Site, Miranda, New South Wales
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, Caboolture, Queensland
  - Pfizer Investigational Site, Kippa-Ring, Queensland
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
- Pfizer Investigational Site, Santiago, RM, Chile
- France (6):
  - Pfizer Investigational Site, Armentières
  - Pfizer Investigational Site, Lorient
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Strasbourg
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
- Pfizer Investigational Site, San Luis Potosí City, San Luis Potosí, Mexico
- Pfizer Investigational Site, Seoul, South Korea
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- United Kingdom (5):
  - Pfizer Investigational Site, Watford, Herts
  - Pfizer Investigational Site, Warminster, Wiltshire
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Luton
  - Pfizer Investigational Site, Northwood, Middlesex

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351019&StudyName=Effect%20of%202-year%20administration%20of%20CP-945%2C598%20on%20weight%20loss%20efficacy%20and%20safety.